CLINICAL TRIAL: NCT01859689
Title: A Phase II Study of Targeted Brachytherapy for Low Risk Prostate Cancer Patients
Brief Title: Internal Radiation Therapy in Treating Patients With Low-Risk Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-003235; NCI-2013-00647 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-04-04; First posted 2013-05-22 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2014-01

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer; Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy; Therapeutics; Radiotherapy, Image-Guided

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (image-guided HDR brachytherapy) (Experimental): Patients undergo 3 fractions of image-guided HDR brachytherapy over 2 days.
  Interventions: Radiation: brachytherapy; Radiation: image-guided radiation therapy; Other: laboratory biomarker analysis

INTERVENTIONS:
Radiation: brachytherapy — Undergo image-guided HDR brachytherapy
  Other Names: low-LET implant therapy; radiation brachytherapy; therapy, low-LET implant
Radiation: image-guided radiation therapy — Undergo image-guided HDR brachytherapy
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well internal radiation therapy works in treating patients with low-risk prostate cancer. Internal radiation uses radioactive material placed directly into or near a tumor to kill tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine long term 5 year prostate specific cancer (PSA) biochemical control using the Phoenix definition of PSA nadir + 2 of targeted hemi-gland brachytherapy.

SECONDARY OBJECTIVES:

I. To assess acute and late toxicity outcomes following targeted brachytherapy according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0.

II. To determine changes from baseline in health-related quality of life indicators using the validated Expanded Prostate Cancer Index Composite (EPIC) questionnaire, International Index of Erectile Function (IIEF) questionnaire, and International Prostate Symptom Score (IPSS) questionnaire.

III. To assess the potential value of multiparametric magnetic resonance imaging, including dynamic contrast enhancement perfusion imaging and diffusion tensor neurovascular tactographic imaging in predicting the development of equivocal disease (ED) following radiation treatment.

OUTLINE:

Patients undergo 3 fractions of image-guided high-dose rate (HDR) brachytherapy over 2 days.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary non-metastatic adenocarcinoma of the prostate
* Unilateral prostate cancer as determined by prostate biopsy
* Less than or equal to 3 positive biopsy cores
* No biopsy core >= 50% positive for cancer
* Karnofsky performance status (KPS) >= 70
* At least a 12 core prostate biopsy; if this was not performed then it will be repeated here at University of California at Los Angeles (UCLA)
* Artemis guided biopsy of any suspicious target lesions as identified on multiparametric (mp)-magnetic resonance imaging (MRI)
* Clinical stage T1c or T2a
* PSA < 10 ng/ml
* Gleason score 3+3=6

Exclusion Criteria:

* Patients who have previously received radiation therapy to the pelvis
* Refusal to sign the informed consent
* Patients who are participating in a concurrent treatment protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Biochemical PSA control using the Phoenix definition of PSA nadir + 2 | 5 years

SECONDARY OUTCOMES:
Grade 3-5 acute toxicity genitourinary (GU) and gastrointestinal (GI) toxicity, graded based on NCI CTCAE v4.0 | 3 months
Grade 3-5 late toxicity GU and GI toxicity, graded based on NCI CTCAE v4.0 | 6 months
Changes in health related quality of life (HR-QOL) as determined by EPIC scores | Up to 24 months
Changes in HR-QOL as determined by IIEF scores | Up to 24 months
Changes in HR-QOL as determined by IPSS scores | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Kamrava, Principal Investigator — Jonsson Comprehensive Cancer Center